CLINICAL TRIAL: NCT04059614
Title: Comparison of High-Flow Nasal Cannula (HFNC) and Conventional Oxygen Therapy (COT) to Diaphragm Function of Post-Upper Abdominal Surgery Patients
Brief Title: Comparison of HFNC and COT to Diaphragm Function of Post-upper Abdominal Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Sidharta K. Manggala, Consultant, Anesthesiologist, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IndonesiaUAnes028
Record Dates: First submitted 2019-06-27; First posted 2019-08-16 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Post Abdominal Surgery
Keywords: HFNC; conventional oxygen; EIT; diaphragm thickness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "High flow nasal cannula (HFNC)" (Active Comparator): "HFNC group: those who receive high-flow nasal cannula therapy
  Interventions: Procedure: HFNC; COT
- conventional oxygen therapy (COT) (Experimental): COT group: those who receive conventional oxygen therapy group
  Interventions: Procedure: HFNC; COT

INTERVENTIONS:
Procedure: HFNC; COT — "HFNC: high-flow nasal cannula therapy COT: conventional oxygen therapy"

SUMMARY:
This study aims to compare diaphragm thickness, air lung distribution, and several clinical and laboratory parameters on post abdominal surgery patients with conventional oxygen therapy vs high-flow nasal cannula

DETAILED DESCRIPTION:
"Approval from Ethical Committee of Faculty of Medicine Universitas Indonesia was acquired prior conducting the study. Subjects were recruited using consecutive sampling method. Subjects underwent upper-abdominal surgery were screened. Eligible and consented subjects were randomized into intervention group (high-flow nasal cannula) and control group (conventional oxygen therapy). Subject and operation characteristics were recorded prior to intervention.

Clinical parameters (vital signs, Borg Score, ICON) were recorded in 10 specific times. diaphragm thickness data using abdominal ultrasonography (USG) and air lung distribution data using Electrical Impedance Tomography were collected in 7 specific times while lactate and blood gas analysis were done 4 times. "

ELIGIBILITY:
Inclusion Criteria:

* patients from 18 - 65 yrs old,
* American Society of Anaesthesia (ASA) status I-III,
* BMI < 30, patent airway,
* Measurement of Exercise Tolerance before Surgery (METS) Score > 4,
* P-POSSUM score <10%,
* agreed to the study

Exclusion Criteria:

* uncooperative subjects,
* DNR (do not resuscitate) patients,
* patients with tracheostomy, pleural effusion, pneumothorax or pulmonary atelectasis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
diaphragm thickness | 2 months
  diaphragm thickness are measured sequentially by abdominal ultrasonography (mm)

SECONDARY OUTCOMES:
electrical impedance tomography (EIT) data | 2 months
  measured data to assess lung ventilation volume and air distribution
partial 02 pressure | 2 months
  partial 02 pressure were collected from arterial blood gas analysis (mmHg)
partial carbondioxyde pressure | 2 months
  partial CO2 pressure were collected from arterial blood gas analysis (mmHg)
ICON | 2 months
  ICON were measured to observe hemodynamic status
lactate | 2 months
  lactate were measured from arterial blood
heart rate | 2 months
  measured from monitor (bpm)
mean arterial pressure | 2 months
  measured from monitor (mmHg)
respiratory rate | 2 months
  bpm

CONTACTS AND LOCATIONS:
Overall Officials: Sidharta K Manggala, Consultant, Principal Investigator — Indonesia University
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Futier E, Paugam-Burtz C, Constantin JM, Pereira B, Jaber S. The OPERA trial - comparison of early nasal high flow oxygen therapy with standard care for prevention of postoperative hypoxemia after abdominal surgery: study protocol for a multicenter randomized controlled trial. Trials. 2013 Oct 18;14:341. doi: 10.1186/1745-6215-14-341. PMID 24138710
- [Result] Futier E, Marret E, Jaber S. Perioperative positive pressure ventilation: an integrated approach to improve pulmonary care. Anesthesiology. 2014 Aug;121(2):400-8. doi: 10.1097/ALN.0000000000000335. No abstract available. PMID 25050494
- [Result] Nishimura M. High-flow nasal cannula oxygen therapy in adults. J Intensive Care. 2015 Mar 31;3(1):15. doi: 10.1186/s40560-015-0084-5. eCollection 2015. PMID 25866645
- [Result] Ni YN, Luo J, Yu H, Liu D, Liang BM, Yao R, Liang ZA. Can high-flow nasal cannula reduce the rate of reintubation in adult patients after extubation? A meta-analysis. BMC Pulm Med. 2017 Nov 17;17(1):142. doi: 10.1186/s12890-017-0491-6. PMID 29149868
- [Result] Zhao H, Wang H, Sun F, Lyu S, An Y. High-flow nasal cannula oxygen therapy is superior to conventional oxygen therapy but not to noninvasive mechanical ventilation on intubation rate: a systematic review and meta-analysis. Crit Care. 2017 Jul 12;21(1):184. doi: 10.1186/s13054-017-1760-8. PMID 28701227
- [Result] Narita M, Tanizawa K, Chin K, Ikai I, Handa T, Oga T, Niimi A, Tsuboi T, Mishima M, Uemoto S, Hatano E. Noninvasive ventilation improves the outcome of pulmonary complications after liver resection. Intern Med. 2010;49(15):1501-7. doi: 10.2169/internalmedicine.49.3375. Epub 2010 Aug 2. PMID 20686280
- [Result] Jaber S, Lescot T, Futier E, Paugam-Burtz C, Seguin P, Ferrandiere M, Lasocki S, Mimoz O, Hengy B, Sannini A, Pottecher J, Abback PS, Riu B, Belafia F, Constantin JM, Masseret E, Beaussier M, Verzilli D, De Jong A, Chanques G, Brochard L, Molinari N; NIVAS Study Group. Effect of Noninvasive Ventilation on Tracheal Reintubation Among Patients With Hypoxemic Respiratory Failure Following Abdominal Surgery: A Randomized Clinical Trial. JAMA. 2016 Apr 5;315(13):1345-53. doi: 10.1001/jama.2016.2706. PMID 26975890
- [Result] Lee BC, Kyoung KH, Kim YH, Hong SK. Non-invasive ventilation for surgical patients with acute respiratory failure. J Korean Surg Soc. 2011 Jun;80(6):390-6. doi: 10.4174/jkss.2011.80.6.390. Epub 2011 Jun 9. PMID 22066065
- [Result] Riera J, Perez P, Cortes J, Roca O, Masclans JR, Rello J. Effect of high-flow nasal cannula and body position on end-expiratory lung volume: a cohort study using electrical impedance tomography. Respir Care. 2013 Apr;58(4):589-96. doi: 10.4187/respcare.02086. PMID 23050520
- [Result] Frerichs I, Amato MB, van Kaam AH, Tingay DG, Zhao Z, Grychtol B, Bodenstein M, Gagnon H, Bohm SH, Teschner E, Stenqvist O, Mauri T, Torsani V, Camporota L, Schibler A, Wolf GK, Gommers D, Leonhardt S, Adler A; TREND study group. Chest electrical impedance tomography examination, data analysis, terminology, clinical use and recommendations: consensus statement of the TRanslational EIT developmeNt stuDy group. Thorax. 2017 Jan;72(1):83-93. doi: 10.1136/thoraxjnl-2016-208357. Epub 2016 Sep 5. PMID 27596161
- [Result] Umbrello M, Formenti P, Longhi D, Galimberti A, Piva I, Pezzi A, Mistraletti G, Marini JJ, Iapichino G. Diaphragm ultrasound as indicator of respiratory effort in critically ill patients undergoing assisted mechanical ventilation: a pilot clinical study. Crit Care. 2015 Apr 13;19(1):161. doi: 10.1186/s13054-015-0894-9. PMID 25886857